CLINICAL TRIAL: NCT04727372
Title: Social Acceptability of COVID-19 Vaccines in Pakistan: Fear and Social Trends
Brief Title: Social Acceptability of COVID-19 Vaccines in Pakistan
Status: Completed | Type: Observational
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Jafir Hussain Shirazi, Lecturer, Islamia University of Bahawalpur
Other Study IDs: Living amongst the fear
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Social Acceptance, Social Anxiety
Keywords: Acceptance; Anxiety; Fear; Social Behavior
MeSH Terms: conditions — Anxiety Disorders; Social Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Islamabad Group: Individuals residing and surveyed in Islamabad
  Interventions: Other: Questionnaire
- Lahore Group: Individuals residing and surveyed in Lahore
  Interventions: Other: Questionnaire
- Faisalabad Group: Individuals residing and surveyed in Faisalabad
  Interventions: Other: Questionnaire
- Bahawalpur Group: Individuals residing and surveyed in Bahawalpur

INTERVENTIONS:
Other: Questionnaire — A structured questionnaire will be served to each participant of study after getting the verbal consent from him for inclusion into the study
  Groups: Faisalabad Group; Islamabad Group; Lahore Group

SUMMARY:
Social settings of Pakistan is unique in the sense that it is composed of multilingual, multicultural and different ethnicities. Also their believes and faiths are so unpredictable. It is therefore observed that this social phenomenon affects the acceptability of new things in this area. Polio vaccination has not worked so well in the past. Iodized salt acceptability has also been criticized in the last decades and is a matter of controversy till now. This behavior has also developed before the commencement of vaccination of COVID-19 in Pakistan, as there are many rumors and fears circulating via social media amongst Pakistan. What will be the acceptance rate for this vaccination, the time will decide.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Cooperative
* Willing to participate in study
* Pakistani citizen

Exclusion Criteria:

* Minors
* non-cooperative/unconconcious
* non-citizen of Pakistan

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All residents of pakistan are eligible to be in included in the study regardless of their geo-location and residencey
Sampling Method: Probability Sample
Enrollment: 986 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Demographics (Age) | Till 23 February 2021
  This is a survey based study in which questionnaire based survey will be conducted. Respondents will be asked about their age, their response will be recorded.
Demographics (Weight) | Till 23 February 2021
  This is a survey based study in which questionnaire based survey will be conducted. Respondents will be asked about their weight and their response will be recorded.
Demographics (Gender) | Till 23 February 2021
  This is a survey based study in which questionnaire based survey will be conducted. Respondents will be asked about their gender and their response will be recorded.
Demographics (Education) | Till 23 February 2021
  This is a survey based study in which questionnaire based survey will be conducted. Respondents will be asked about their level of education and their response will be recorded.
Demographics (Family set up) | Till 23 February 2021
  This is a survey based study in which questionnaire based survey will be conducted. Respondents will be asked about their family set i.e. joint family or separate family and their response will be recorded.
Demographics (Residence) | Till 23 February 2021
  This is a survey based study in which questionnaire based survey will be conducted. Respondents will be asked about their residence i.e. either in rural area or living in city and their response will be recorded.
Attitude, knowledge and behavior about COVID-19 Vaccine and its acceptance or rejection | Till 23 February 2021
  As this is a survey based study in which questionnaire based survey will be conducted. Respondents will be asked about vaccines, knowledge about vaccines, about corona vaccine specifically, about efficacy of vaccines, about efficacy of COVID-19 vaccine. about acceptance or rejection of vaccine, if they will not have a shot of vaccine then reasons, if they will have shots then reason for vaccination. if they are fear off vaccines then their reasons

SECONDARY OUTCOMES:
Correlation of Age with a particular behavior | Till the end of February 2021
  Statistical Analysis of raw data about age will be computed. Various age groups will be classified and arranged. Frequencies of these age groups will be calculated and will be analyzed about any relationship with a particular behavior about vaccination.
Correlation of Weight with a particular behavior | Till 23 February 2021
  Statistical Analysis of raw data about age will be computed. Various age groups will be classified and arranged. Frequencies of these age groups will be calculated and will be analyzed about any relationship with a particular behavior about vaccination.
Correlation of Gender with a particular behavior | Till 23 February 2021
  Statistical Analysis of raw data about age will be computed. Various age groups will be classified and arranged. Frequencies of these age groups will be calculated and will be analyzed about any relationship with a particular behavior about vaccination.
Correlation of Education level with a particular behavior | Till 23 February 2021
  Statistical Analysis of raw data about age will be computed. Various age groups will be classified and arranged. Frequencies of these age groups will be calculated and will be analyzed about any relationship with a particular behavior about vaccination.
Correlation of Family set up with a particular behavior | Till 23 February 2021
  Statistical Analysis of raw data about age will be computed. Various age groups will be classified and arranged. Frequencies of these age groups will be calculated and will be analyzed about any relationship with a particular behavior about vaccination.
Correlation of Residence with a particular behavior | Till 23 February 2021
  Statistical Analysis of raw data about age will be computed. Various age groups will be classified and arranged. Frequencies of these age groups will be calculated and will be analyzed about any relationship with a particular behavior about vaccination.
Respondents Attitude, knowledge and behavior about COVID-19 Vaccine and its acceptance or rejection | Till 23 February 2021
  Statistical Analysis of raw data about age will be computed. Various age groups will be classified and arranged. Frequencies of these age groups will be calculated and will be analyzed about any relationship with a particular behavior about vaccination. t-Test will be applied to observe any statistically significant difference between different co-variates

CONTACTS AND LOCATIONS:
Overall Officials: Jafir Shirazi, PhD, Principal Investigator — The Islamia University of Bahawalpur; Anam Sharmeen, M. Phil, Study Director — The Islamia University of Bahawalpur; Asfa Akbar, M. Phil, Study Chair — The Islamia University of Bahawalpur; Fouzia Akbar, M.Phil, Study Chair — The Islamia University of Bahawalpur
Locations (4):
- Pakistan (4):
  - Islamabad City, Islamabad, Capital Territory
  - Bahawalpur Rural and Urban Areas, Bahawalpur, Punjab Province
  - Faisalabad city, Faisalābad, Punjab Province
  - Lahore City, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No